CLINICAL TRIAL: NCT00499603
Title: Open Label Randomized Clinical Trial of Standard Neoadjuvant Chemotherapy (Paclitaxel Followed by FEC) Versus the Combination of Paclitaxel and RAD001 Followed by FEC in Women With Triple Receptor-Negative Breast Cancer (CRAD001C24101)
Brief Title: Paclitaxel Followed by FEC Versus Paclitaxel and RAD001 Followed by FEC In Women With Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0790; NCI-2012-01514 (Registry Identifier: NCI CTRP); 1K23CA121994-1 (Other Grant/Funding Number: NCI); 1K23CA121994 (NIH)
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; ER negative; PR negative; HER2neu negative; Tumor Triple Negative Receptors; Paclitaxel; Taxol; RAD001; FEC; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Epirubicin; Cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Fluorouracil; Epirubicin; Cyclophosphamide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel + FEC (Experimental): Paclitaxel 80 mg/m^2 intravenously (IV) on day 1(+/- 2 days) of each week, followed by four cycles of combination 5-Fluorouracil at 500 mg/m^2, Epirubicin at 100 mg/m^2 and Cyclophosphamide at 500 mg/m^2 (FEC) on day 1 every 3 weeks (+/- 7 days).
  Interventions: Drug: Paclitaxel; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide
- Paclitaxel + RAD001 + FEC (Experimental): Paclitaxel + RAD001 Followed by FEC (5-Fluorouracil + Epirubicin + Cyclophosphamide)
  Interventions: Drug: Paclitaxel; Drug: 5-Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: RAD001

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m^2 by vein once weekly over 1 hour on day 1(+/- 2 days) each week for 3 weeks and for 12 cycles.
  Other Names: Taxol
Drug: 5-Fluorouracil — 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Epirubicin — 100 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
Drug: Cyclophosphamide — 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Other Names: Cytoxan®; Neosar®
Drug: RAD001 — 30 mg by mouth weekly on Days 1, 8, & 15 for 12 cycles.
  Arms: Paclitaxel + RAD001 + FEC

SUMMARY:
The goal of this clinical research is to learn if RAD001 given in combination with chemotherapy will turn off the signaling pathway (a chain of information that tells cancer cells to grow quickly) and make the chemotherapies given on this study more effective.

Primary Objective

· To determine if the addition of an mTOR inhibitor to standard neoadjuvant chemotherapy in patients with triple receptor-negative breast cancer causes molecular changes (inhibition/activation) of the PI3K/PTEN/AKT pathway.

Secondary Objectives

* To evaluate pathologic complete response (pCR) rates for each treatment group.
* To evaluate the relationship between pCR and the molecular changes (inhibition/activation) of the PI13K/PTEN/AKT pathway in each treatment group.
* To evaluate overall response rates (ORR) for each treatment group.
* To assess the toxicity of both regimens and to evaluate the relationship of toxicities with PI3K/PTEN/AKT pathway status.

DETAILED DESCRIPTION:
RAD001 is a new drug that was designed to block proteins that are important in the development and growth of cancer. It may also stop the growth of new blood vessels that help tumor growth, resulting in cell death.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam. Blood (about 6 tablespoons) will be drawn for routine tests and to test for the amount of fat in the blood. You will have a chest x-ray, bone scan and a 2-D echocardiogram (a test to evaluate the pumping function of the heart). You will have a computed tomography (CT) scan of the chest and abdomen (stomach area). Women who are able to have children must have a negative blood (about 1 tablespoon) pregnancy test.

You will have a mammogram and an ultrasound of the breast and armpit to record tumor size. As part of this study, you will have a fine needle biopsy of the breast tumor to test for the signaling pathway. You will receive a separate consent form for the mammogram, ultrasound, and biopsy and these procedures will be discussed with you in more detail. The fine needle biopsy is a procedure that would not be performed if you were not on this study.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. You will have an equal chance of being assigned to either group.

If you are assigned to Group 1, you will receive paclitaxel once a week through a needle in your vein over 1 hour. You will have a total of 12 treatments. Before each treatment, you may also receive drugs to help prevent or reduce your risk of side effects from paclitaxel.

If you are assigned to Group 2, you will receive paclitaxel and RAD001. You will receive paclitaxel once a week through a needle in your vein over 1 hour. You will have a total of 12 treatments. Before each treatment, you may also receive drugs to help prevent or reduce your risk of side effects from paclitaxel. You will take RAD001, by mouth, on each day you receive paclitaxel. You should take RAD001 on an empty stomach or after a light meal. Pills will not be taken out of their package until the staff is ready for you to take them, since they can be damaged by light or humidity.

Participants in both groups will have blood (about 2 tablespoons) drawn for routine tests before each weekly dose of chemotherapy.

You will have a second fine needle biopsy 2 days after starting treatment. This will be done to check to see if the signaling pathway has been affected.

After your 12 weeks of treatment with paclitaxel or paclitaxel and RAD001, you will have an ultrasound and if tumor is visible, a fine needle biopsy to check to see if the signaling pathway has been affected.

After the 12 week treatment with either paclitaxel or paclitaxel and RAD001, you will begin treatment with 5-fluorouracil, epirubicin, and cyclophosphamide. This drug combination is called FEC. You will receive FEC through needle in your vein (over 1 hour) once every 3 weeks. You will have 4 treatments (12 weeks total). Before each treatment, you may also receive drugs to help prevent or reduce your risk of side effects from FEC.

Once you have finished treatment with FEC, you will have a mammogram and ultrasound to check the status of the disease. This mammogram and ultrasound will also be used by the doctor to decide whether to remove all or part of the breast and/or nearby lymph nodes during surgery.

You will then have surgery to remove all or part of the breast that has the tumor. If there are signs that the lymph nodes in the armpit contain cancer, these lymph nodes will also be removed. You will receive a separate consent form for these procedures and your doctor will discuss them in more detail. If available, a portion of left over tumor tissue will be collected to check to see if the signaling pathway has been affected.

You will be considered "off study" once you have had surgery. You will be taken off study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Paclitaxel, 5-fluorouracil, cyclophosphamide, and epirubicin are all FDA approved and commercially available. RAD001 is not FDA approved or commercially available. It has been authorized for use in research only. Up to 50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic confirmation of invasive ER/PR and HER2/neu-negative breast carcinoma. Immunohistochemistry (IHC) must be used for ER/PR evaluation and IHC or FISH for determination of HER2/neu. ER/PR will be considered negative if equal or lower than 5% IHC staining and HER2/neu will be considered negative if IHC of 0% or negative FISH.
2. Patients must have intact primary tumors.
3. Age equal or greater than 18 years
4. Patients should have stage IIA (T1N1) to IIIC non inflammatory breast cancer.
5. Patients with bilateral breast cancers are eligible.
6. Patients should have a Karnofsky performance scale of =/> 70%.
7. Patients must have clinically measurable disease to be treated in the neoadjuvant setting. This includes patients with a non-palpable primary tumor who have histologically proven lymph node involvement that is clinically palpable and measurable by ultrasound.
8. Patients should have adequate bone marrow function, as defined by peripheral granulocyte count of >/= 1500/mm3, and a platelet count >/= 100000/ mm3.
9. Patients must have adequate liver function with a bilirubin within normal laboratory values. Alkaline phosphatase and transaminases (ALT and AST) may be up to 1.5 x upper limit of normal (ULN) of the institution.
10. Patients should have adequate renal function with creatinine levels 2.0 mg/dL or lower
11. Patients should have a normal left ventricular ejection fraction of =/> 50%.
12. Negative serum pregnancy test for a woman of childbearing potential.
13. Women of childbearing potential (WOCBP) must use a reliable and appropriate contraceptive method during the study and 6 months after chemotherapy is completed. WOCBP are women who are not menopausal for 12 months or had no previous surgical sterilization.
14. Patients must agree to have study biopsies.
15. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.
16. Hemoglobin 9.0 gm/dL or higher

Exclusion Criteria:

1. Patients whose tumors express ER, PR or HER2/neu gene amplification.
2. Patients with a history of other invasive malignancies diagnosed and treated within the previous 5 years, except non-melanoma skin cancer and non-invasive cervical cancer
3. Patients with an organ allograft or other history of immune compromise
4. Prior exposure to mTOR inhibitors
5. Hypersensitivity to rapamycin or other similar compounds
6. Prior treatment with any investigational drug within the preceding 4 weeks
7. Chronic treatment with systemic steroids or another immunosuppressive agent
8. A known history of HIV seropositivity
9. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
10. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin defined as 1 mg a day).
11. Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration)
12. Patients with a pre-existing peripheral neuropathy > grade 1
13. Patients taking medications metabolized by the CYP3A4 subfamily will not be included in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2017-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gonzalez-Angulo AM, Akcakanat A, Liu S, Green MC, Murray JL, Chen H, Palla SL, Koenig KB, Brewster AM, Valero V, Ibrahim NK, Moulder-Thompson S, Litton JK, Tarco E, Moore J, Flores P, Crawford D, Dryden MJ, Symmans WF, Sahin A, Giordano SH, Pusztai L, Do KA, Mills GB, Hortobagyi GN, Meric-Bernstam F. Open-label randomized clinical trial of standard neoadjuvant chemotherapy with paclitaxel followed by FEC versus the combination of paclitaxel and everolimus followed by FEC in women with triple receptor-negative breast cancerdagger. Ann Oncol. 2014 Jun;25(6):1122-7. doi: 10.1093/annonc/mdu124. Epub 2014 Mar 24. PMID 24669015
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with triple negative breast cancer who were seen in the Breast Medical Oncology clinic of the MD Anderson Cancer Center were enrolled in the study prior to surgery from August 16, 2007 to September 14, 2010.
Pre-assignment Details: Sixty-two (62) participants were registered but only fifty (50) were randomized. Nine patients failed the screening process, two patients withdrew consent, and one patient was discontinued due to therapy interruption for greater than 21 days.
Groups:
- Paclitaxel + FEC: Paclitaxel 80 mg/m^2 intravenously (IV) on day 1(+/- 2 days) of each week, followed by four cycles of combination 5-Fluorouracil at 500 mg/m^2, Epirubicin at 100 mg/m^2 and Cyclophosphamide at 500 mg/m^2 (FEC) on day 1 every 3 weeks (+/- 7 days).
  5-Fluorouracil : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Paclitaxel : 80 mg/m^2 by vein once weekly over 1 hour on day 1(+/- 2 days) each week for 3 weeks and for 12 cycles.
  Cyclophosphamide: 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Epirubicin : 100 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
- Paclitaxel + RAD001 + FEC: Paclitaxel + RAD001 Followed by FEC (5-Fluorouracil + Epirubicin + Cyclophosphamide)
  5-Fluorouracil : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Paclitaxel : 80 mg/m^2 by vein once weekly over 1 hour on day 1(+/- 2 days) each week for 3 weeks and for 12 cycles.
  RAD001 : 30 mg by mouth weekly on Days 1, 8, & 15 for 12 cycles.
  Cyclophosphamide: 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Epirubicin : 100 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
Period: Overall Study
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC
Started | 27 | 23
Completed | 27 | 22
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel + FEC: Paclitaxel 80 mg/m^2 intravenously (IV) on day 1(+/- 2 days) of each week, followed by four cycles of combination 5-Fluorouracil at 500 mg/m^2, Epirubicin at 100 mg/m^2 and Cyclophosphamide at 500 mg/m^2 (FEC) on day 1 every 3 weeks (+/- 7 days).
  5-Fluorouracil : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Paclitaxel : 80 mg/m^2 by vein once weekly over 1 hour on day 1(+/- 2 days) each week for 3 weeks and for 12 cycles.
  Cyclophosphamide : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Epirubicin : 100 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
- Paclitaxel + RAD001 + FEC: Paclitaxel + RAD001 Followed by FEC (5-Fluorouracil + Epirubicin + Cyclophosphamide)
  5-Fluorouracil : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Paclitaxel : 80 mg/m^2 by vein once weekly over 1 hour on day 1(+/- 2 days) each week for 3 weeks and for 12 cycles.
  RAD001 : 30 mg by mouth weekly on Days 1, 8, & 15 for 12 cycles.
  Cyclophosphamide : 500 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
  Epirubicin : 100 mg/m^2 by vein on day 1 every 3 weeks (+/- 7 days) for 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Median (Full Range); unit: years] | 52 [30 to 65] | 46 [32 to 75] | 48 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50
Cancer Clinical Stage [Number; unit: participants] — Clinical staging describes the extent or severity of a person's cancer where T1, T2, T3, T4 define the size and/or extent of the primary tumor with the higher numbers indicating more extensive disease.
  participants
    T1 | 4 | 3 | 7
    T2 | 18 | 17 | 35
    T3 | 4 | 1 | 5
    T4 | 1 | 1 | 2
    Unknown or Not Reported | 0 | 1 | 1
Regional Lymph Node Stage [Number; unit: Participants] — Regional lymph node staging illustrates the amount of cancer spread to nearby lymph nodes, notations are NX: Regional lymph nodes cannot be evaluated; N0: No regional lymph node involvement; N1, N2, N3: Degree of regional lymph node involvement (number and location of lymph nodes)
  Participants
    N0 | 8 | 6 | 14
    N1 | 10 | 7 | 17
    N2 | 4 | 2 | 6
    Nx | 5 | 7 | 12
    Unknown or Not Reported | 0 | 1 | 1
Breast Cancer Stage [Number; unit: Participants] — Participants staged using histologically confirmed disease stages Stage IIA, IIB and IIIA, IIIB, IIIC per the American Joint Committee on Cancer (AJCC) sixth edition for breast cancer.
  Participants
    IIA | 8 | 8 | 16
    IIB | 8 | 6 | 14
    IIIA | 4 | 2 | 6
    IIIB | 2 | 0 | 2
    IIIC | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With Inhibition of PI3K/PTEN/AKT Pathway at 48 Hours
Description: Number of participants with inhibition of the PI3K/PTEN/AKT pathway at 48 hours after the start of treatment, regardless of the status of the pathway at the time of randomization. Molecular changes (inhibition/activation) of the PI3K/PTEN/AKT pathway evaluated using reverse phase protein arrays (RPPA) where fine-needle aspirations (FNAs) from the primary breast cancer obtained pretreatment, and at 48 hours. Bioinformatics cluster analysis of arrays used to define molecular changes as inhibition or activation where pathways called 'active' with presence of 2 or more phosphorilated pathway proteins (pAKT, pmTOR, pGSK3, pS6K1, pS6), and 'inhibited' with one or none phosphorilated pathway proteins present.
Time Frame: 48 hours after start of treatment
Population: Participants were randomly assigned 1:1 to receive T-FEC or TR-FEC using a balanced block design stratified by disease stage and menopausal status. One participant in Arm 2 started treatment but had untolerable side effects and was taken off the study and thus was considered inevaluable.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC
Number analyzed (Participants) | 27 | 22
participants | 27 | 22

2. Secondary Outcome: Participant Responses Per Treatment Arm at 12 Weeks
Description: Radiographic criteria of response based on regional ultrasound examination (decrease in size of the primary tumor and/or fatty replacement in regional lymph nodes), and includes partial response and complete response. A decrease in size of the product of the two largest dimensions =/> 50% considered a partial response (PR), and a complete disappearance of the primary tumor by physical exam and or ultrasound and normalization of the lymph nodes by ultrasound will be considered a complete clinical response (CR). Stable Disease (SD) is carcinoma neither decreasing nor increasing in extent or severity, and Progression of disease (PD) defined as 30% increase in size primary tumor and/or lymph nodes on physical exam and/or ultrasound.
Time Frame: 12 weeks
Population: Participants who did not complete the entire 12 week of paclitaxel +/- RAD001 or the entire 4 cycles of FEC are evaluable for response.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC
Number analyzed (Participants) | 27 | 23
participants
  CR | 3 | 0
  PR | 5 | 11
  SD | 16 | 11
  PD | 3 | 1

3. Secondary Outcome: Participant Responses Per Treatment Arm at 24 Weeks
Description: as for outcome 2
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC
Number analyzed (Participants) | 27 | 23
participants
  CR | 4 | 2
  PR | 16 | 11
  SD | 7 | 7
  PD | 0 | 3

ADVERSE EVENTS:
Time Frame: 3 years and 9 months
Description: Serious Adverse Events reported include Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 and Grade 4 combined within each arm. Other Adverse Events were not assessed.
Arm/Group | Paclitaxel + FEC | Paclitaxel + RAD001 + FEC
Serious Adverse Events (participants affected / at risk) | 27/27 | 23/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + FEC (N=27) | Paclitaxel + RAD001 + FEC (N=23)
Fatigue (Blood and lymphatic system disorders) | 2 (2) | 4 (4) — Combined CTCAE Grade 3 & 4 events
GI Disturbaces (Gastrointestinal disorders) | 5 (5) | 6 (6)
Neuropathy (Vascular disorders) | 1 (1) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 11 (11) | 12 (12)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Increased leukocytes (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nail changes (General disorders) | 0 (0) | 1 (1)
Edema of extremities (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hypokalemia (Investigations) | 0 (0) | 1 (1)
Syncope (General disorders) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No